CLINICAL TRIAL: NCT04910477
Title: Comparative Effects of Nebulized Dexmedetomidine Versus Neostigmine / Atropine in Treating Postdural Puncture Headache After Cesarean Section: A Double Blind Randomized Clinical Trial
Brief Title: Nebulized Dexmedetomidine Versus Neostigmine/Atropine in Postdural Puncture Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300608
Record Dates: First submitted 2021-05-25; First posted 2021-06-02 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Dexmedetomidine; Neostigmine; Atropine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine (Experimental): Group D (patients will receive ultrasonic nebulization of dexmedetomidine (1 mg/kg diluted in 4 mL saline) twice daily for three days.
  Interventions: Drug: Dexmedetomidine
- Neostigmine/atropine (Experimental): Group N (patients will receive nebulization of 20 µ/kg neostigmine and 10 µ/kg atropine mixed in 4 ml) twice daily for three days.
  Interventions: Drug: Neostigmine/atropine
- Saline placebo (Placebo Comparator): Group S (patients will receive nebulization of saline placebo in 4 ml)twice daily for three days.
  Interventions: Other: Saline placebo

INTERVENTIONS:
Drug: Dexmedetomidine — ultrasonic nebulization of dexmedetomidine (1 mg/kg diluted in 4 mL saline) twice daily for three days.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Neostigmine/atropine — nebulization of 20 µ/kg neostigmine and 10 µ/kg atropine mixed in 4 ml) twice daily for three days.
  Arms: Neostigmine/atropine
Other: Saline placebo — nebulization of saline placebo in 4 ml) twice daily for three days.
  Other Names: Normal saline
  Arms: Saline placebo

SUMMARY:
In our study, we will compare a new route of nebulization for effectiveness between dexmedetomidine, neostigmine/atropine and saline placebo for females complained of postdural puncture headache (PDPH) after cesarean section.

DETAILED DESCRIPTION:
A written informed consent will be taken from the patients. The study will involve female adults (age 18-40years) of American society of anesthesiologists (ASA) I-II who are listed for elective cesarean section under spinal anesthesia and suffer from postoperative postdural puncture headache (PDPH). Patients will be assigned randomly to three groups (30 subjects each) after PDPH diagnosis was established. First 90 patients developed PDPH will be assessed for study eligibility.

Group D (patients will receive ultrasonic nebulization of dexmedetomidine (1 mg/kg diluted in 4 mL saline) twice daily for three days. Group N (patients will receive nebulization of 20 µ/kg neostigmine and 10 µ/kg atropine mixed in 4 ml) twice daily for three days. Group S (patients will receive nebulization of saline placebo in 4 ml) twice daily for three days.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of postdural puncture headache (PDPH) after elective cesarean section under spinal anesthesia.

Exclusion Criteria:

* Hypersensitivity of dexmedetomidine, neostigmine or atropine
* Overactive thyroid gland
* Myasthenia gravis
* Closed angle glaucoma
* High blood pressure and coronary artery disease.
* withdrawal of consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female suffering from PDPH after cesarean section
Enrollment: 90 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
visual analog scale score (VAS) ≤3 within 72 hour. | 3 days
  change in visual analog scale score (VAS )for the assessment of the degree of headache (with 0 representing no headache and 10 cm representing the worst imaginable headache). a visual analog scale score ≤3 within 72 hour after intervention will be recorded.

SECONDARY OUTCOMES:
Need for Epidural blood patch | Day 4
  Epidural blood patch will be done in failed study drugs, traditional treatment and taking consent from patients after 72h from intervention
Occurence of neck stiffness | 3 days
  If there is occurance of neck stiffness after start of PDPH

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, Principal Investigator — Omar makram
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided